CLINICAL TRIAL: NCT04585009
Title: A Randomised Double-blind, Placebo Controlled, Single Ascending and Repeat Dose, First Time in Human Study in Healthy Participants and Stable Asthmatics to Assess Safety, Tolerability and Pharmacokinetics of GSK3923868 Inhalation Powder
Brief Title: Safety, Tolerability and Pharmacokinetics of GSK3923868 Inhalation Powder in Healthy Participants and Stable Asthmatics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 213497
Record Dates: First submitted 2020-10-09; First posted 2020-10-14 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: First time in human; Stable asthmatics; GSK3923868; Inhalation powder; Phosphatidylinositol 4-kinase beta
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Part A will be a single ascending dose escalation study consisting of two sequential cross-over cohorts (Cohorts 1 and 2) in healthy participants. Part B is a repeat dose study consisting of two parallel cohorts (Cohort 3 and 4) in healthy participants. Part C is a repeat dose study consisting of one cohort (Cohort 5) in participants with asthma.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Cohort1:GSK3923868 50 micrograms (mcg)/ Placebo/ 250mcg (Experimental): Healthy participants will receive single ascending doses of GSK3923868 or placebo in the planned treatment sequence: GSK3923868 50 mcg/Placebo/250 mcg in treatment periods 1, 2 and 3 respectively. There will be at least 10 days of wash-out period between doses for each participant.
  Interventions: Drug: GSK3923868; Drug: Matching placebo; Device: Monodose RS01
- Cohort 1:GSK3923868 50 mcg/ 100 mcg/ Placebo (Experimental): Healthy participants will receive single ascending doses of GSK3923868 or placebo in the planned treatment sequence: GSK3923868 50 mcg/100 mcg/Placebo in treatment periods 1, 2 and 3 respectively. There will be at least 10 days of wash-out period between doses for each participant.
  Interventions: Drug: GSK3923868; Drug: Matching placebo; Device: Monodose RS01
- Cohort 1:GSK3923868 50mcg/ 100mcg/ 250mcg (Experimental): Healthy participants will receive single ascending doses of GSK3923868 in the planned treatment sequence: GSK3923868 50 mcg/100 mcg/250 mcg in treatment periods 1, 2 and 3 respectively. There will be at least 10 days of wash-out period between doses for each participant.
  Interventions: Drug: GSK3923868; Device: Monodose RS01
- Cohort 1:Placebo / GSK3923868 100 mcg/ GSK3923868 250 mcg (Experimental): Healthy participants will receive single ascending doses of GSK3923868 or placebo in the planned treatment sequence: Placebo/GSK3923868 100 mcg/GSK3923868 250 mcg in treatment periods 1, 2 and 3 respectively. There will be at least 10 days of wash-out period between doses for each participant.
  Interventions: Drug: GSK3923868; Drug: Matching placebo; Device: Monodose RS01
- Cohort 2:Placebo / GSK3923868 1000 mcg/ GSK3923868 3000 mcg (Experimental): Healthy participants will receive single ascending doses of GSK3923868 or placebo in the planned treatment sequence: Placebo/GSK3923868 1000 mcg/GSK3923868 3000 mcg. There will be at least 10 days of wash-out period between doses for each participant.
  Interventions: Drug: GSK3923868; Drug: Matching placebo; Device: Monodose RS01
- Cohort 2:GSK3923868 500 mcg/ Placebo/ 3000 mcg (Experimental): Healthy participants will receive single ascending doses of GSK3923868 or placebo in the planned treatment sequence: GSK3923868 500 mcg/Placebo/3000 mcg. There will be at least 10 days of wash-out period between doses for each participant.
  Interventions: Drug: GSK3923868; Drug: Matching placebo; Device: Monodose RS01
- Cohort 2:GSK3923868 500 mcg/ 1000 mcg/ Placebo (Experimental): Healthy participants will receive single ascending doses of GSK3923868 or placebo in the planned treatment sequence: GSK3923868 500 mcg/1000 mcg/Placebo. There will be at least 10 days of wash-out period between doses for each participant.
  Interventions: Drug: GSK3923868; Drug: Matching placebo; Device: Monodose RS01
- Cohort 2:GSK3923868 500mcg/ 1000mcg/ 3000mcg (Experimental): Healthy participants will receive single ascending doses of GSK3923868 in the planned treatment sequence: GSK3923868 500 mcg/1000 mcg/3000 mcg. There will be at least 10 days of wash-out period between doses for each participant.
  Interventions: Drug: GSK3923868; Device: Monodose RS01
- Cohort 3: Participants receivings repeated doses of GSK3923868 (Experimental): Healthy participants will receive planned repeat doses of 3000 mcg (six capsules) GSK3923868 daily for 14 days
  Interventions: Drug: GSK3923868; Device: Monodose RS01
- Cohort 4: Participants receiving repeat doses of GSK3923868 (Experimental): Healthy participants will receive planned repeat doses of 3000 mcg (six capsules) GSK3923868 daily for 14 days
  Interventions: Drug: GSK3923868; Device: Monodose RS01
- Cohort 5: Participants receiving repeat doses of GSK3923868 (Experimental): Participants with stable asthma will receive a planned repeat dosing of 3000 mcg (six capsules) GSK3923868 daily for 7 days
  Interventions: Drug: GSK3923868; Device: Monodose RS01

INTERVENTIONS:
Drug: GSK3923868 — GSK3923868 will be available as capsules containing inhalation powder blend to be delivered via Monodose RS01 device.
Drug: Matching placebo — Placebo to match GSK3923868 will be available as capsule containing inhalation powder to be delivered via Monodose RS01 device.
  Arms: Cohort 1:GSK3923868 50 mcg/ 100 mcg/ Placebo; Cohort 1:Placebo / GSK3923868 100 mcg/ GSK3923868 250 mcg; Cohort 2:GSK3923868 500 mcg/ 1000 mcg/ Placebo; Cohort 2:GSK3923868 500 mcg/ Placebo/ 3000 mcg; Cohort 2:Placebo / GSK3923868 1000 mcg/ GSK3923868 3000 mcg; Cohort1:GSK3923868 50 micrograms (mcg)/ Placebo/ 250mcg
Device: Monodose RS01 — Participants will receive GSK3923868 and placebo as capsules containing inhalation powder blend to be delivered via Monodose RS01 device.

SUMMARY:
This is a first time in human (FTIH) study designed to evaluate the safety, tolerability and pharmacokinetic (PK) profile of single and repeat doses of GSK3923868 inhalation powder in both healthy participants and asthmatics. This is a 3-part, randomized, double blind, placebo controlled study of GSK3923868, administered as an inhalation powder blend (GSK3923868 capsules for inhalation) via Mono-dose inhaler in healthy participants (Parts A and B) and in participants with asthma (Part C). The duration of study participation for each part A, B and C will be 11, 9 and 8 weeks, respectively.

ELIGIBILITY:
Inclusion Criteria: For Parts A and B

* Between 18 and 50 years of age inclusive, at the time of signing the informed consent.
* Participants who are generally healthy as determined by medical evaluation based on screening medical history, physical examination, vital signs, ECG assessment, pulmonary function testing, laboratory tests and cardiac monitoring.
* Body weight at least 50.0 kilograms (kg) (110 pounds [lbs]) and body mass index (BMI) within the range 18.5 to 32.0 kilograms per meter square (kg/m^2) (inclusive).
* Male Participants: A male participant is eligible to participate if they agree to the following during the intervention period and for at least 10 days after the last dose of study intervention: Refrain from donating sperm. Plus either be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remaining abstinent OR must agree to use contraception as detailed below when having sexual intercourse with a woman of childbearing potential who is not currently pregnant: Agree to use a male condom AND female partner to use an additional highly effective contraceptive method with a failure rate of < 1 percent per year. The participant should also be advised of the benefit for a female partner as a condom may break or leak.
* Female Participants: A female participant is eligible to participate if she is not pregnant or breastfeeding and is a woman of non-childbearing potential (WONCBP).
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and protocol.

Inclusion Criteria: Part C

* Between 18 and 50 years of age inclusive, at the time of signing the informed consent.
* Participants who are otherwise healthy (other than the acceptable condition of asthma and other mild atopic diseases, including allergic rhinitis and atopic dermatitis) as determined by medical evaluation based on screening medical history, physical examination, vital signs, ECG assessment, pulmonary function testing, laboratory tests and cardiac monitoring.
* A physician diagnosis of asthma (as defined by the Global Initiative for Asthma [GINA], 2020 guidelines) at least 6 months before screening. The reason for diagnosis of asthma should be documented in the participant's source data, including relevant history.
* A screening pre-bronchodilator FEV1 >= 65 percent predicted normal value.
* Positive bronchodilator reversibility test defined as an increase in FEV1 of > 12 percent and > 200 milliliter (mL) from Baseline, 10 to 15 minutes after administration of 400 micrograms (μg) salbutamol (or equivalent).
* Participants with maintained control of their asthma using the permitted medications: short-acting beta agonist (SABA) use only (n=8 participants) and regular treatment with inhaled corticosteroid (ICS) or ICS/long-acting beta agonist (LABA) (including use of Leukotriene Receptor Agonist [LTRA]) (n=8 participants).
* Body weight at least 50.0 kg (110 lbs) and BMI within the range 18.5 to 32.0 kg/m^2 (inclusive).
* Male Participants: A male participant is eligible to participate if they agree to the following during the intervention period and for at least 10 days after the last dose of study intervention: Refrain from donating sperm plus either be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remaining abstinent OR must agree to use contraception as detailed below when having sexual intercourse with a woman of childbearing potential who is not currently pregnant: Agree to use a male condom AND female partner to use an additional highly effective contraceptive method with a failure rate of < 1 percent per year. The participant should also be advised of the benefit for a female partner as a condom may break or leak.
* Female Participants: A female participant is eligible to participate if she is not pregnant or breastfeeding and is a WONCBP.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria: Part A and B

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data.
* Alanine transaminase (ALT) and Aspartate Aminotransferase (AST) above upper limit of normal (ULN).
* Total Bilirubin above ULN (isolated bilirubin above ULN is acceptable if total bilirubin is fractionated and direct bilirubin <35 percent).
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QTcF > 450 milliseconds (msec) at screening visit based on the average of triplicate ECGs.
* Screening ECG measurements meets the following criteria for exclusion: heart rate: males- <45 or > 100 beats per minute (bpm); females- <50 or > 100 bpm; PR interval: <120 or >220 msec; QRS duration: <70 or >120 msec; QTcF: >450 msec.
* Medical history of cardiac arrhythmias or cardiac disease or a family or personal history of long QT syndrome.
* Evidence of previous myocardial infarction (does not include ST segment changes associated with re-polarization).
* Signs and symptoms suggestive of COVID-19.
* Past or intended use of over-the-counter or prescription medication, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days before the first dose of study intervention, unless in the opinion of the Investigator and the GlaxoSmithKline (GSK) Medical Monitor, the medication will not interfere with the study procedures or compromise participant safety.
* Participation in this study would result in loss of blood or blood products in excess of 500 milliliter (mL) within 56 days.
* Exposure to more than 4 new chemical entities within 12 months before the first dosing day.
* Current enrolment or past participation in a clinical trial and has received an investigational product within the following time period before the first dosing day in this study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* FEV1 and FVC is < 80 percent predicted normal value.
* Presence of hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to first dose of study intervention.
* Positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention.
* Positive hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study intervention.
* Positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* Positive test for COVID-19 infection.
* Current or history of drug abuse.
* Any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular (AV) block [2nd degree or higher], Wolff-Parkinson-White (WPW) syndrome).
* Sinus Pauses > 3 seconds.
* Any significant arrhythmia which, in the opinion of the Investigator or GSK Medical monitor, will interfere with the safety for the individual participant.
* Non-sustained or sustained ventricular tachycardia (with more than 3 consecutive ventricular ectopic beats).
* Regular alcohol consumption within 6 months prior to the study defined as: an average weekly intake of > 14 units for both males and females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Current or previous use of tobacco- or nicotine-containing products (e.g. cigarettes, nicotine patches or electronic devices) within 6 months before screening and/or have a smoking pack history of > 5 pack years.
* Positive breath carbon monoxide test indicative of recent smoking at screening or each in-house admission to the clinical research unit.
* Sensitivity to any of the study interventions, or components thereof (including lactose and magnesium stearate [MgSt]), or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.
* Participants with known COVID-19 positive contacts in the past 14 days.

Exclusion criteria: Part C

* Any asthma exacerbation requiring systemic corticosteroids within 8 weeks of screening, or that resulted in overnight hospitalization requiring additional treatment for asthma within 3 months of screening.
* A history of life-threatening asthma, defined as an any asthma episode that required admission to a high-dependency or intensive therapy unit.
* Significant pulmonary diseases, other than asthma, including (but not limited to): pneumonia previously requiring hospital admission, bronchiectasis, pulmonary fibrosis, bronchopulmonary dysplasia, chronic bronchitis, emphysema, chronic obstructive pulmonary disease, or other significant respiratory abnormalities.
* ALT and AST above ULN.
* Bilirubin above ULN (isolated bilirubin above ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QTcF > 450 msec at screening visit based on the average of triplicate ECGs.
* Signs and symptoms suggestive of COVID-19.
* Past or intended use of over-the-counter or prescription medication, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days before the first dose of study intervention, unless in the opinion of the Investigator and the GSK Medical Monitor, the medication will not interfere with the study procedures or compromise participant safety.
* Participation in this study would result in loss of blood or blood products in excess of 500 mL within 56 days.
* Exposure to more than 4 new chemical entities within 12 months before the first dosing day.
* Current enrolment or past participation in a clinical trial and has received an investigational product within the following time period before the first dosing day in this study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Presence of HBsAg at screening or within 3 months prior to first dose of study intervention.
* Positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention.
* Positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study intervention.
* Positive pre-study drug/alcohol screen.
* Positive HIV antibody test.
* Positive test for COVID-19 infection.
* Current or history of drug abuse.
* Regular alcohol consumption within 6 months prior to the study defined as: an average weekly intake of > 14 units for males and females. One unit is equivalent to 8 g of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Current or previous use of tobacco- or nicotine-containing products (e.g. cigarettes, nicotine patches or electronic devices) within 6 months before screening and/or have a smoking pack history of > 5 pack years.
* Positive breath carbon monoxide test indicative of recent smoking at screening or each in-house admission to the clinical research unit.
* Sensitivity to any of the study interventions, or components thereof (including lactose and MgSt), or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.
* Participants with known COVID-19 positive contacts in the past 14 days.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a three-part study with single dose escalation in Part A and repeat dose in Part B and C. Part A and B was conducted in healthy volunteers and Part C was conducted in participants with asthma.
Pre-assignment Details: A total of 56 participants (28 in Part A ,17 in Part B and 11 in Part C) were enrolled in this study. This study was conducted at a single center in the United Kingdom.
Groups:
- Cohort 1: GSK3923868 50 Micrograms (mcg)/ Placebo/ 250mcg: Healthy participants received single ascending doses of GSK3923868, or placebo matched to GSK3923868 on Day 1 in the planned treatment sequence: GSK3923868 50 mcg/Placebo/250 mcg in treatment periods 1, 2 and 3 respectively. There was a washout of at least 10 days after Treatment Periods 1 and 2. Participants were followed up for 7 to 14 days after last dose in Treatment Period 3.
- Cohort 1: GSK3923868 50 mcg/ 100 mcg/ Placebo: Healthy participants received single ascending doses of GSK3923868, or placebo matched to GSK3923868 on Day 1 in the planned treatment sequence: GSK3923868 50 mcg/100 mcg/Placebo in treatment periods 1, 2 and 3 respectively. There was a washout of at least 10 days after Treatment Periods 1 and 2. Participants were followed up for 7 to 14 days after last dose in Treatment Period 3.
- Cohort 1: GSK3923868 50mcg/ 100mcg/ 250mcg: Healthy participants received single ascending doses of GSK3923868 on Day 1 in the planned treatment sequence: GSK3923868 50 mcg/100 mcg/250 mcg in treatment periods 1, 2 and 3 respectively. There was a washout of at least 10 days after Treatment Periods 1 and 2. Participants were followed up for 7 to 14 days after last dose in Treatment Period 3.
- Cohort 1: Placebo / GSK3923868 100 mcg/ 250 mcg: Healthy participants received single ascending doses of GSK3923868, or placebo matched to GSK3923868 on Day1 in the planned treatment sequence: Placebo/GSK3923868 100 mcg/GSK3923868 250 mcg in treatment periods 1, 2 and 3 respectively. There was a washout of at least 10 days after Treatment Periods 1 and 2. Participants were followed up for 7 to 14 days after last dose in Treatment Period 3.
- Cohort 2: Placebo / GSK3923868 1000 mcg/ 3000 mcg: Healthy participants received single ascending doses of GSK3923868, or placebo matched to GSK3923868 on Day 1 in the planned treatment sequence: Placebo/GSK3923868 1000 mcg/GSK3923868 3000 mcg in treatment periods 4, 5 and 6 respectively. There was a washout of at least 10 days after Treatment Periods 4 and 5. Participants were followed up for 7 to 14 days after last dose in Treatment Period 6.
- Cohort 2: GSK3923868 500 mcg/ Placebo/ 3000 mcg: Healthy participants received single ascending doses of GSK3923868, or placebo matched to GSK3923868 on Day 1 in the planned treatment sequence: GSK3923868 500 mcg/Placebo/3000 mcg in treatment periods 4, 5 and 6 respectively. There was a washout of at least 10 days after Treatment Periods 4 and 5. Participants were followed up for 7 to 14 days after last dose in Treatment Period 6.
- Cohort 2: GSK3923868 500 mcg/ 1000 mcg/ Placebo: Healthy participants received single ascending doses of GSK3923868, or placebo matched to GSK3923868 on Day 1 in the planned treatment sequence: GSK3923868 500 mcg/1000 mcg/Placebo in treatment periods 4, 5 and 6 respectively. There was a washout of at least 10 days after Treatment Periods 4 and 5. Participants were followed up for 7 to 14 days after last dose in Treatment Period 6.
- Cohort 2: GSK3923868 500mcg/ 1000mcg/ 3000mcg: Healthy participants received single ascending doses of GSK3923868 on Day 1 in the planned treatment sequence: GSK3923868 500 mcg/1000 mcg/3000 mcg in treatment periods 4, 5 and 6 respectively. There was a washout of at least 10 days after Treatment Periods 4 and 5. Participants were followed up for 7 to 14 days after last dose in Treatment Period 6.
- Cohort 3 and 4: Placebo: Healthy participants received placebo matched to GSK3923868 daily for 14 days. Participants were followed up for 7 to 14 days post last dose of the study treatment.
- Cohort 3 and 4: GSK3923868 3000mcg: Healthy participants received planned repeat doses of 3000 mcg GSK3923868 daily for 14 days. Participants were followed up for 7 to 14 days post last dose of the study treatment.
- Cohort 5: Placebo: Participants with stable asthma received placebo matched to GSK3923868 daily for 7 days. Participants were followed up for 7 to 14 days post last dose of the study treatment.
- Cohort 5: GSK3923868 3000mcg: Participants with stable asthma received a planned repeat dosing of 3000 mcg GSK3923868 daily for 7 days. Participants were followed up for 7 to 14 days post last dose of the study treatment.
Period: PartA, Cohort1, Treatment Period1(Day1)
Arm/Group | Cohort 1: GSK3923868 50 Micrograms (mcg)/ Placebo/ 250mcg | Cohort 1: GSK3923868 50 mcg/ 100 mcg/ Placebo | Cohort 1: GSK3923868 50mcg/ 100mcg/ 250mcg | Cohort 1: Placebo / GSK3923868 100 mcg/ 250 mcg | Cohort 2: Placebo / GSK3923868 1000 mcg/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ Placebo/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ 1000 mcg/ Placebo | Cohort 2: GSK3923868 500mcg/ 1000mcg/ 3000mcg | Cohort 3 and 4: Placebo | Cohort 3 and 4: GSK3923868 3000mcg | Cohort 5: Placebo | Cohort 5: GSK3923868 3000mcg
Started | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort1: Washout Period1 (10Days)
Arm/Group | Cohort 1: GSK3923868 50 Micrograms (mcg)/ Placebo/ 250mcg | Cohort 1: GSK3923868 50 mcg/ 100 mcg/ Placebo | Cohort 1: GSK3923868 50mcg/ 100mcg/ 250mcg | Cohort 1: Placebo / GSK3923868 100 mcg/ 250 mcg | Cohort 2: Placebo / GSK3923868 1000 mcg/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ Placebo/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ 1000 mcg/ Placebo | Cohort 2: GSK3923868 500mcg/ 1000mcg/ 3000mcg | Cohort 3 and 4: Placebo | Cohort 3 and 4: GSK3923868 3000mcg | Cohort 5: Placebo | Cohort 5: GSK3923868 3000mcg
Started | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PartA, Cohort1,Treatment Period2(Day1)
Arm/Group | Cohort 1: GSK3923868 50 Micrograms (mcg)/ Placebo/ 250mcg | Cohort 1: GSK3923868 50 mcg/ 100 mcg/ Placebo | Cohort 1: GSK3923868 50mcg/ 100mcg/ 250mcg | Cohort 1: Placebo / GSK3923868 100 mcg/ 250 mcg | Cohort 2: Placebo / GSK3923868 1000 mcg/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ Placebo/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ 1000 mcg/ Placebo | Cohort 2: GSK3923868 500mcg/ 1000mcg/ 3000mcg | Cohort 3 and 4: Placebo | Cohort 3 and 4: GSK3923868 3000mcg | Cohort 5: Placebo | Cohort 5: GSK3923868 3000mcg
Started | 3 (One new participant enrolled and dosed.) | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort1: Washout Period2(10 Days)
Arm/Group | Cohort 1: GSK3923868 50 Micrograms (mcg)/ Placebo/ 250mcg | Cohort 1: GSK3923868 50 mcg/ 100 mcg/ Placebo | Cohort 1: GSK3923868 50mcg/ 100mcg/ 250mcg | Cohort 1: Placebo / GSK3923868 100 mcg/ 250 mcg | Cohort 2: Placebo / GSK3923868 1000 mcg/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ Placebo/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ 1000 mcg/ Placebo | Cohort 2: GSK3923868 500mcg/ 1000mcg/ 3000mcg | Cohort 3 and 4: Placebo | Cohort 3 and 4: GSK3923868 3000mcg | Cohort 5: Placebo | Cohort 5: GSK3923868 3000mcg
Started | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PartA, Cohort1, Treatment Period3(Day1)
Arm/Group | Cohort 1: GSK3923868 50 Micrograms (mcg)/ Placebo/ 250mcg | Cohort 1: GSK3923868 50 mcg/ 100 mcg/ Placebo | Cohort 1: GSK3923868 50mcg/ 100mcg/ 250mcg | Cohort 1: Placebo / GSK3923868 100 mcg/ 250 mcg | Cohort 2: Placebo / GSK3923868 1000 mcg/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ Placebo/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ 1000 mcg/ Placebo | Cohort 2: GSK3923868 500mcg/ 1000mcg/ 3000mcg | Cohort 3 and 4: Placebo | Cohort 3 and 4: GSK3923868 3000mcg | Cohort 5: Placebo | Cohort 5: GSK3923868 3000mcg
Started | 3 (One new participant enrolled and dosed.) | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PartA, Cohort2: Treatment Period4(Day1)
Arm/Group | Cohort 1: GSK3923868 50 Micrograms (mcg)/ Placebo/ 250mcg | Cohort 1: GSK3923868 50 mcg/ 100 mcg/ Placebo | Cohort 1: GSK3923868 50mcg/ 100mcg/ 250mcg | Cohort 1: Placebo / GSK3923868 100 mcg/ 250 mcg | Cohort 2: Placebo / GSK3923868 1000 mcg/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ Placebo/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ 1000 mcg/ Placebo | Cohort 2: GSK3923868 500mcg/ 1000mcg/ 3000mcg | Cohort 3 and 4: Placebo | Cohort 3 and 4: GSK3923868 3000mcg | Cohort 5: Placebo | Cohort 5: GSK3923868 3000mcg
Started | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 2 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Cohort2: Washout Period1 (10 Days)
Arm/Group | Cohort 1: GSK3923868 50 Micrograms (mcg)/ Placebo/ 250mcg | Cohort 1: GSK3923868 50 mcg/ 100 mcg/ Placebo | Cohort 1: GSK3923868 50mcg/ 100mcg/ 250mcg | Cohort 1: Placebo / GSK3923868 100 mcg/ 250 mcg | Cohort 2: Placebo / GSK3923868 1000 mcg/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ Placebo/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ 1000 mcg/ Placebo | Cohort 2: GSK3923868 500mcg/ 1000mcg/ 3000mcg | Cohort 3 and 4: Placebo | Cohort 3 and 4: GSK3923868 3000mcg | Cohort 5: Placebo | Cohort 5: GSK3923868 3000mcg
Started | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 2 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 2 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PartA, Cohort2: Treatment Period5(Day1)
Arm/Group | Cohort 1: GSK3923868 50 Micrograms (mcg)/ Placebo/ 250mcg | Cohort 1: GSK3923868 50 mcg/ 100 mcg/ Placebo | Cohort 1: GSK3923868 50mcg/ 100mcg/ 250mcg | Cohort 1: Placebo / GSK3923868 100 mcg/ 250 mcg | Cohort 2: Placebo / GSK3923868 1000 mcg/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ Placebo/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ 1000 mcg/ Placebo | Cohort 2: GSK3923868 500mcg/ 1000mcg/ 3000mcg | Cohort 3 and 4: Placebo | Cohort 3 and 4: GSK3923868 3000mcg | Cohort 5: Placebo | Cohort 5: GSK3923868 3000mcg
Started | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 (One new participant enrolled and dosed.) | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort2: Washout Period2 (10 Days)
Arm/Group | Cohort 1: GSK3923868 50 Micrograms (mcg)/ Placebo/ 250mcg | Cohort 1: GSK3923868 50 mcg/ 100 mcg/ Placebo | Cohort 1: GSK3923868 50mcg/ 100mcg/ 250mcg | Cohort 1: Placebo / GSK3923868 100 mcg/ 250 mcg | Cohort 2: Placebo / GSK3923868 1000 mcg/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ Placebo/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ 1000 mcg/ Placebo | Cohort 2: GSK3923868 500mcg/ 1000mcg/ 3000mcg | Cohort 3 and 4: Placebo | Cohort 3 and 4: GSK3923868 3000mcg | Cohort 5: Placebo | Cohort 5: GSK3923868 3000mcg
Started | 0 | 0 | 0 | 0 | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PartA, Cohort2: Treatment Period6(Day1)
Arm/Group | Cohort 1: GSK3923868 50 Micrograms (mcg)/ Placebo/ 250mcg | Cohort 1: GSK3923868 50 mcg/ 100 mcg/ Placebo | Cohort 1: GSK3923868 50mcg/ 100mcg/ 250mcg | Cohort 1: Placebo / GSK3923868 100 mcg/ 250 mcg | Cohort 2: Placebo / GSK3923868 1000 mcg/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ Placebo/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ 1000 mcg/ Placebo | Cohort 2: GSK3923868 500mcg/ 1000mcg/ 3000mcg | Cohort 3 and 4: Placebo | Cohort 3 and 4: GSK3923868 3000mcg | Cohort 5: Placebo | Cohort 5: GSK3923868 3000mcg
Started | 0 | 0 | 0 | 0 | 3 (One new participant enrolled and dosed.) | 3 | 3 | 3 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B, Cohorts 3 & 4 (Days 1 to 14)
Arm/Group | Cohort 1: GSK3923868 50 Micrograms (mcg)/ Placebo/ 250mcg | Cohort 1: GSK3923868 50 mcg/ 100 mcg/ Placebo | Cohort 1: GSK3923868 50mcg/ 100mcg/ 250mcg | Cohort 1: Placebo / GSK3923868 100 mcg/ 250 mcg | Cohort 2: Placebo / GSK3923868 1000 mcg/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ Placebo/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ 1000 mcg/ Placebo | Cohort 2: GSK3923868 500mcg/ 1000mcg/ 3000mcg | Cohort 3 and 4: Placebo | Cohort 3 and 4: GSK3923868 3000mcg | Cohort 5: Placebo | Cohort 5: GSK3923868 3000mcg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 13 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 12 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Part C, Cohort 5 (Days 1 to 7)
Arm/Group | Cohort 1: GSK3923868 50 Micrograms (mcg)/ Placebo/ 250mcg | Cohort 1: GSK3923868 50 mcg/ 100 mcg/ Placebo | Cohort 1: GSK3923868 50mcg/ 100mcg/ 250mcg | Cohort 1: Placebo / GSK3923868 100 mcg/ 250 mcg | Cohort 2: Placebo / GSK3923868 1000 mcg/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ Placebo/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ 1000 mcg/ Placebo | Cohort 2: GSK3923868 500mcg/ 1000mcg/ 3000mcg | Cohort 3 and 4: Placebo | Cohort 3 and 4: GSK3923868 3000mcg | Cohort 5: Placebo | Cohort 5: GSK3923868 3000mcg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: GSK3923868 50 Micrograms (mcg)/ Placebo/ 250mcg | Cohort 1: GSK3923868 50 mcg/ 100 mcg/ Placebo | Cohort 1: GSK3923868 50mcg/ 100mcg/ 250mcg | Cohort 1: Placebo / GSK3923868 100 mcg/ 250 mcg | Cohort 2: Placebo / GSK3923868 1000 mcg/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ Placebo/ 3000 mcg | Cohort 2: GSK3923868 500 mcg/ 1000 mcg/ Placebo | Cohort 2: GSK3923868 500mcg/ 1000mcg/ 3000mcg | Cohort 3 and 4: Placebo | Cohort 3 and 4: GSK3923868 3000mcg | Cohort 5: Placebo | Cohort 5: GSK3923868 3000mcg | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 4 | 3 | 3 | 4 | 4 | 13 | 3 | 8 | 56
Age, Customized [Count of Participants; unit: Participants]
  <=18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  19-64 | 5 | 3 | 3 | 3 | 4 | 3 | 3 | 4 | 4 | 13 | 3 | 8 | 56
  >=65 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 5 | 3 | 3 | 3 | 4 | 3 | 3 | 4 | 4 | 13 | 3 | 8 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4
  BLACK OR AFRICAN AMERICAN | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 7
  WHITE | 3 | 3 | 2 | 2 | 3 | 2 | 3 | 4 | 2 | 11 | 2 | 7 | 44
  MIXED RACE | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part A, Cohort-1: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AEs and SAEs were collected. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is any untoward medical occurrence that, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity and/or can result in death. Number of participants with AEs and SAEs assessed in Part A, Cohort-1 from the start of dosing and post-dose washout period (10 days) after treatment periods was reported.
Time Frame: Up to Day 43
Population: The analysis was performed on the safety set that includes all randomized participants who received at least 1 dose of study intervention. Participants were analyzed according to the treatment they received.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Placebo: Healthy participants received a single dose (SD) of placebo matched to GSK3923868 in one of the 3 treatment periods. A washout period of at least 10 days was maintained between treatment periods. Participants were followed up for 7 to 14 days post last dose of the study treatment.
- Cohort 1: GSK3923868 50 mcg: Healthy participants received a SD of GSK3923868 50 mcg in one of the 3 treatment periods. A washout period of at least 10 days was maintained between treatment periods. Participants were followed up for 7 to 14 days post last dose of the study treatment.
- Cohort 1: GSK3923868 100 mcg: Healthy participants received a SD of GSK3923868 100 mcg in one of the 3 treatment periods. A washout period of at least 10 days was maintained between treatment periods. Participants were followed up for 7 to 14 days post last dose of the study treatment.
- Cohort 1: GSK3923868 250mcg: Healthy participants received a SD of GSK3923868 250 mcg in one of the 3 treatment periods. A washout period of at least 10 days was maintained between treatment periods. Participants were followed up for 7 to 14 days post last dose of the study treatment.
Arm/Group | Cohort 1: Placebo | Cohort 1: GSK3923868 50 mcg | Cohort 1: GSK3923868 100 mcg | Cohort 1: GSK3923868 250mcg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  AEs | 3 | 3 | 3 | 6
  SAEs | 0 | 0 | 0 | 0

2. Primary Outcome: Part A, Cohort 2: Number of Participants With AEs and SAEs
Description: AEs and SAEs were collected. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is any untoward medical occurrence that, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity and/or can result in death. Number of participants with AEs and SAEs assessed in Part A, Cohort-2 from the start of dosing and post-dose washout period (10 days) after treatment periods was reported.
Time Frame: Up to Day 43
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Placebo: Healthy participants received a SD of placebo matched to GSK3923868 in one of the 3 treatment periods. A washout period of at least 10 days was maintained between treatment periods. Participants were followed up for 7 to 14 days post last dose of the study treatment.
- Cohort 2: GSK3923868 500 mcg: Healthy participants received a SD of GSK3923868 500 mcg in one of the 3 treatment periods. A washout period of at least 10 days was maintained between treatment periods. Participants were followed up for 7 to 14 days post last dose of the study treatment.
- Cohort 2: GSK3923868 1000 mcg: Healthy participants received a SD of GSK3923868 1000 mcg in one of the 3 treatment periods. A washout period of at least 10 days was maintained between treatment periods. Participants were followed up for 7 to 14 days post last dose of the study treatment.
- Cohort 2: GSK3923868 3000mcg: Healthy participants received a SD of GSK3923868 3000 mcg in one of the 3 treatment periods. A washout period of at least 10 days was maintained between treatment periods. Participants were followed up for 7 to 14 days post last dose of the study treatment.
Arm/Group | Cohort 2: Placebo | Cohort 2: GSK3923868 500 mcg | Cohort 2: GSK3923868 1000 mcg | Cohort 2: GSK3923868 3000mcg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  AEs | 5 | 5 | 5 | 3
  SAEs | 0 | 0 | 0 | 0

3. Primary Outcome: Part B: Number of Participants With AEs and SAEs
Description: AEs and SAEs were collected. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is any untoward medical occurrence that, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity and/or can result in death. Number of participants with AEs and SAEs assessed in Part B, Cohort-3 and 4 (repeat dose) of the study were reported. Part B assessed repeat doses of study drug across two parallel cohorts (Cohorts 3 and 4).
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 3 and 4: Placebo: Healthy participants received placebo daily for 14 days. Participants were followed up for 7 to 14 days post last dose of the study treatment.
Arm/Group | Cohort 3 and 4: Placebo | Cohort 3 and 4: GSK3923868 3000mcg
Number analyzed (Participants) | 4 | 13
Participants
  AEs | 4 | 12
  SAEs | 0 | 0

4. Primary Outcome: Part C: Number of Participants With AEs and SAEs
Description: AEs and SAEs were collected. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is any untoward medical occurrence that, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity and/or can result in death. Number of participants with AEs and SAEs assessed in Part C, Cohort-5 (repeat dose) of the study were reported.
Time Frame: Up to Day 21
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 5: Placebo | Cohort 5: GSK3923868 3000mcg
Number analyzed (Participants) | 3 | 8
Participants
  AEs | 3 | 8
  SAEs | 0 | 0

5. Primary Outcome: Part A, Cohort-1: Number of Participants With Clinically Significant Changes in Clinical Chemistry and Hematology Laboratory Parameters
Description: The laboratory (lab) measurements included Clinical chemistry and hematology. The parameters evaluated were hemoglobin, leukocytes, lymphocytes/leukocytes, neutrophils/leukocytes, platelets, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, red blood cells, reticulocytes, Alanine Aminotransferase (ALT), Albumin, Alkaline Phosphatase, Aspartate Aminotransferase, Bilirubin, Calcium Corrected for Albumin, Creatinine, Glucose, Potassium and Sodium. Number of participants with clinically significant changes from baseline in clinical chemistry and hematology were reported. Clinical significance was determined by the investigator.
Time Frame: From start of the treatment (Day 1) to Day 2 in each treatment period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: GSK3923868 50 mcg | Cohort 1: GSK3923868 100 mcg | Cohort 1: GSK3923868 250mcg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Clinical Chemistry | 0 | 0 | 0 | 0
  Hematology | 0 | 0 | 0 | 0

6. Primary Outcome: Part A, Cohort-2: Number of Participants With Clinically Significant Changes in Clinical Chemistry and Hematology Lab Parameters
Description: as for outcome 5
Time Frame: From start of the treatment (Day 1) to Day 2 in each treatment period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Placebo | Cohort 2: GSK3923868 500 mcg | Cohort 2: GSK3923868 1000 mcg | Cohort 2: GSK3923868 3000mcg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Clinical Chemistry | 0 | 0 | 0 | 0
  Hematology | 0 | 0 | 0 | 0

7. Primary Outcome: Part B: Number of Participants With Clinically Significant Changes in Clinical Chemistry and Hematology Lab Parameters
Description: The laboratory (lab) measurements included Clinical chemistry and hematology. The parameters evaluated were hemoglobin, leukocytes, lymphocytes/leukocytes, neutrophils/leukocytes, platelets, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, red blood cells, reticulocytes, Alanine Aminotransferase (ALT), Albumin, Alkaline Phosphatase, Aspartate Aminotransferase, Bilirubin, Calcium Corrected for Albumin, Creatinine, Glucose, Potassium and Sodium. Part B assessed repeat doses of study drug across two parallel cohorts (Cohorts 3 and 4). Number of participants with clinically significant changes from baseline in clinical chemistry and hematology were reported. Clinical significance was determined by the investigator.
Time Frame: From start of the treatment (Day 1) to Day 18
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3 and 4: Placebo | Cohort 3 and 4: GSK3923868 3000mcg
Number analyzed (Participants) | 4 | 13
Participants
  Clinical Chemistry | 1 | 0
  Hematology | 0 | 0

8. Primary Outcome: Part C: Number of Participants With Clinically Significant Changes in Clinical Chemistry and Hematology Lab Parameters
Description: as for outcome 5
Time Frame: From start of the treatment (Day 1) to Day 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 5: Placebo | Cohort 5: GSK3923868 3000mcg
Number analyzed (Participants) | 3 | 8
Participants
  Clinical Chemistry | 1 | 1
  Hematology | 0 | 0

9. Primary Outcome: Part A, Cohort-1: Number of Participants With Clinically Significant Changes in Vital Signs and 12-Lead Electrocardiogram (ECG) Findings
Description: Vital signs included systolic and diastolic blood pressure, pulse and respiratory rate and were measured with the participant in semi-supine position after 5 minutes rest. Temperature was also measured as a vital sign but did not require positioning or rest prior to measuring. Twelve-lead electrocardiogram were performed in a semi-supine position using an ECG machine that automatically calculates the heart rate and measures PR interval, QRS duration, QT and corrected QT intervals (QTc) intervals. Number of participants with clinically significant changes in parameters for cohort-1 were reported. Clinical significance was determined by the investigator.
Time Frame: From start of the treatment (Day 1) to Day 2 in each treatment period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Placebo: Healthy participants received a single dose (SD) of placebo in one of the 3 treatment periods. A washout period of at least 10 days was maintained between treatment periods. Participants were followed up for 7 to 14 days post last dose of the study treatment.
Arm/Group | Cohort 1: Placebo | Cohort 1: GSK3923868 50 mcg | Cohort 1: GSK3923868 100 mcg | Cohort 1: GSK3923868 250mcg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Vital Signs | 0 | 0 | 0 | 0
  12-Lead ECG | 0 | 0 | 0 | 0

10. Primary Outcome: Part A, Cohort-2: Number of Participants With Clinically Significant Changes in Vital Signs and 12-Lead ECG Findings
Description: Vital signs included systolic and diastolic blood pressure, pulse and respiratory rate and were measured with the participant in semi-supine position after 5 minutes rest. Temperature was also measured as a vital sign but did not require positioning or rest prior to measuring. Twelve-lead electrocardiogram were performed in a semi-supine position using an ECG machine that automatically calculates the heart rate and measures PR interval, QRS duration, QT and corrected QT intervals (QTc) intervals. Number of participants with clinically significant changes in parameters for cohort-2 were reported. Clinical significance was determined by the investigator.
Time Frame: From start of the treatment (Day 1) to Day 2 in each treatment period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Placebo: Healthy participants received a single dose (SD) of placebo matched to GSK3923868 in one of the 3 treatment periods. A washout period of at least 10 days was maintained between treatment periods. Participants were followed up for 7 to 14 days post last dose of the study treatment.
Arm/Group | Cohort 2: Placebo | Cohort 2: GSK3923868 500 mcg | Cohort 2: GSK3923868 1000 mcg | Cohort 2: GSK3923868 3000mcg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Vital Signs | 0 | 0 | 0 | 0
  12-Lead ECG | 0 | 0 | 0 | 0

11. Primary Outcome: Part B: Number of Participants With Clinically Significant Changes in Vital Signs and 12-Lead ECG Findings
Description: Vital signs included systolic and diastolic blood pressure, pulse and respiratory rate and were measured with the participant in semi-supine position after 5 minutes rest. Temperature was also measured as a vital sign but did not require positioning or rest prior to measuring. Twelve-lead electrocardiogram were performed in a semi-supine position using an ECG machine that automatically calculates the heart rate and measures PR interval, QRS duration, QT and corrected QT intervals (QTc) intervals. Part B assessed repeat doses of study drug across two parallel cohorts (Cohorts 3 and 4). Number of participants with clinically significant changes in parameters were reported. Clinical significance was determined by the investigator.
Time Frame: From start of the treatment (Day 1) to Day 18
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3 and 4: Placebo | Cohort 3 and 4: GSK3923868 3000mcg
Number analyzed (Participants) | 4 | 13
Participants
  Vital Signs | 1 | 6
  12-Lead ECG | 0 | 0

12. Primary Outcome: Part C: Number of Participants With Clinically Significant Changes in Vital Signs and 12-Lead ECG Findings
Description: Vital signs included systolic and diastolic blood pressure, pulse and respiratory rate and were measured with the participant in semi-supine position after 5 minutes rest. Temperature was also measured as a vital sign but did not require positioning or rest prior to measuring. Twelve-lead electrocardiogram were performed in a semi-supine position using an ECG machine that automatically calculates the heart rate and measures PR interval, QRS duration, QT and corrected QT intervals (QTc) intervals. Number of participants with clinically significant changes in parameters for cohort-5 were reported. Clinical significance was determined by the investigator.
Time Frame: From start of the treatment (Day 1) to Day 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 5: Placebo | Cohort 5: GSK3923868 3000mcg
Number analyzed (Participants) | 3 | 8
Participants
  Vital Signs | 0 | 0
  12-Lead ECG | 0 | 0

13. Primary Outcome: Part A, Cohort-1: Number of Participants With Clinically Significant Changes in Spirometry Measurements
Description: Spirometry included forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) for lung function assessment. Number of participants with clinically significant changes in parameters were reported. Clinical significance was determined by the investigator.
Time Frame: From start of the treatment (Day 1) to Day 2 in each treatment period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: GSK3923868 50 mcg | Cohort 1: GSK3923868 100 mcg | Cohort 1: GSK3923868 250mcg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 0 | 0 | 0 | 0

14. Primary Outcome: Part A, Cohort-2: Number of Participants With Clinically Significant Changes in Spirometry Measurements
Description: as for outcome 13
Time Frame: From start of the treatment (Day 1) to Day 2 in each treatment period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Placebo: Healthy participants received a SD of placebo in one of the 3 treatment periods. A washout period of at least 10 days was maintained between treatment periods. Participants were followed up for 7 to 14 days post last dose of the study treatment.
Arm/Group | Cohort 2: Placebo | Cohort 2: GSK3923868 500 mcg | Cohort 2: GSK3923868 1000 mcg | Cohort 2: GSK3923868 3000mcg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 0 | 0 | 0 | 0

15. Primary Outcome: Part B: Number of Participants With Clinically Significant Changes in Spirometry Measurements
Description: as for outcome 13
Time Frame: From start of the treatment (Day 1) up to Day 18
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3 and 4: Placebo | Cohort 3 and 4: GSK3923868 3000mcg
Number analyzed (Participants) | 4 | 13
Participants | 0 | 0

16. Primary Outcome: Part C: Number of Participants With Clinically Significant Changes in Spirometry Measurements
Description: as for outcome 13
Time Frame: From start of the treatment (Day 1) to Day 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 5: Placebo | Cohort 5: GSK3923868 3000mcg
Number analyzed (Participants) | 3 | 8
Participants | 0 | 0

17. Secondary Outcome: Part A, Cohort 1 and 2: Area Under the Plasma GSK3923868 Concentration Versus Time Curve From Time Zero to Last Quantifiable Concentration (AUC[0-t])
Description: Blood samples were collected for measurement of plasma concentrations of GSK3923868. Area under the concentration-time curve from time zero to the time of the last quantifiable concentration values were reported. Single ascending doses of GSK3923868 were assessed in 2 sequential crossover cohorts (Cohorts 1 and 2) of healthy participants, each with up to 3 treatment periods.
Time Frame: Up to Day 2 in each treatment period
Population: The analysis was performed on the Pharmacokinetic (PK) Set that includes all randomized participants who received at least 1 dose of study intervention and had at least 1 non-missing PK assessment (Non-quantifiable [NQ] values were to be considered as non-missing values). Participants were analyzed according to the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*Picograms Per Milliliter (h*pg/mL)
Groups:
- Cohort 1: GSK3923868 50 mcg: Healthy participants received a SD of GSK3923868 50 mcg in one of the 3 treatment periods. A washout period of at least 10 days was maintained between treatment periods.
- Cohort 1: GSK3923868 100 mcg: Healthy participants received a SD of GSK3923868 100 mcg in one of the 3 treatment periods. A washout period of at least 10 days was maintained between treatment periods.
- Cohort 1: GSK3923868 250mcg: Healthy participants received a SD of GSK3923868 250 mcg in one of the 3 treatment periods. A washout period of at least 10 days was maintained between treatment periods.
- Cohort 2: GSK3923868 500 mcg: Healthy participants received a SD of GSK3923868 500 mcg in one of the 3 treatment periods. A washout period of at least 10 days was maintained between treatment periods.
- Cohort 2: GSK3923868 1000 mcg: Healthy participants received a SD of GSK3923868 1000 mcg in one of the 3 treatment periods. A washout period of at least 10 days was maintained between treatment periods.
- Cohort 2: GSK3923868 3000mcg: Healthy participants received a SD of GSK3923868 3000 mcg in one of the 3 treatment periods. A washout period of at least 10 days was maintained between treatment periods.
Arm/Group | Cohort 1: GSK3923868 50 mcg | Cohort 1: GSK3923868 100 mcg | Cohort 1: GSK3923868 250mcg | Cohort 2: GSK3923868 500 mcg | Cohort 2: GSK3923868 1000 mcg | Cohort 2: GSK3923868 3000mcg
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9
Hour*Picograms Per Milliliter (h*pg/mL) | 1774.65 (48.78) | 3810.3 (39.08) | 8111.1 (33.37) | 22550.14 (24.76) | 49756.36 (22.85) | 144519.79 (24.37)

18. Secondary Outcome: Part A, Cohort 1 and 2: Area Under the Plasma GSK3923868 Concentration Versus Time Curve From Time Zero to Infinity (AUC [0-inf])
Description: Blood samples were collected for measurement of plasma concentrations of GSK3923868. Area under the concentration-time curve from time zero extrapolated to infinite time values were reported.
Time Frame: Up to Day 2 in each treatment period
Population: The analysis was performed on the PK Set that includes all randomized participants who received at least 1 dose of study intervention and had at least 1 non-missing PK assessment (NQ values were to be considered as non-missing values). Participants were analyzed according to the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Groups:
- Cohort 1: GSK3923868 50 mcg: Healthy participants received a SD of GSK3923868 50 mcg in one of the 3 treatment periods. A washout of at least 10 days was maintained between treatment periods.
- Cohort 1: GSK3923868 100 mcg: Healthy participants received a SD of GSK3923868 100 mcg in one of the 3 treatment periods. A washout of at least 10 days was maintained between treatment periods.
- Cohort 1: GSK3923868 250mcg: Healthy participants received a SD of GSK3923868 250 mcg in one of the 3 treatment periods. A washout of at least 10 days was maintained between treatment periods.
- Cohort 2: GSK3923868 500 mcg: Healthy participants received a SD of GSK3923868 500 mcg in one of the 3 treatment periods. A washout of at least 10 days was maintained between treatment periods.
- Cohort 2: GSK3923868 1000 mcg: Healthy participants received a SD of GSK3923868 1000 mcg in one of the 3 treatment periods. A washout of at least 10 days was maintained between treatment periods.
- Cohort 2: GSK3923868 3000mcg: Healthy participants received a SD of GSK3923868 3000 mcg in one of the 3 treatment periods. A washout of at least 10 days was maintained between treatment periods.
Arm/Group | Cohort 1: GSK3923868 50 mcg | Cohort 1: GSK3923868 100 mcg | Cohort 1: GSK3923868 250mcg | Cohort 2: GSK3923868 500 mcg | Cohort 2: GSK3923868 1000 mcg | Cohort 2: GSK3923868 3000mcg
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9
h*pg/mL | 1964.21 (50.59) | 4125.22 (40.59) | 8656.56 (34.71) | 22941.62 (24.69) | 50504.33 (22.89) | 146453.53 (24.53)

19. Secondary Outcome: Part A, Cohort 1 and 2: Maximum Observed GSK3923868 Plasma Concentration (Cmax)
Description: Cmax was defined as the maximum concentration of drug GSK3923868 in plasma. Blood samples were collected for measurement of plasma concentrations of GSK3923868 for PK analysis.
Time Frame: Up to Day 2 in each treatment period
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms Per Milliliter (pg/mL)
Arm/Group | Cohort 1: GSK3923868 50 mcg | Cohort 1: GSK3923868 100 mcg | Cohort 1: GSK3923868 250mcg | Cohort 2: GSK3923868 500 mcg | Cohort 2: GSK3923868 1000 mcg | Cohort 2: GSK3923868 3000mcg
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9
Picograms Per Milliliter (pg/mL) | 370.84 (37.29) | 772.49 (29.19) | 1811.8 (27.96) | 4284.89 (23.49) | 9583.02 (25.61) | 30985.12 (26.09)

20. Secondary Outcome: Part A, Cohort 1 and 2: Time to Maximum Observed Plasma Drug Concentration (Tmax)
Description: Tmax was defined as time required to achieve Cmax for drug GSK3923868 in plasma. Blood samples were collected for measurement of plasma concentrations of GSK3923868 for PK analysis.
Time Frame: Up to Day 2 in each treatment period
Population: as for outcome 18
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Cohort 1: GSK3923868 50 mcg | Cohort 1: GSK3923868 100 mcg | Cohort 1: GSK3923868 250mcg | Cohort 2: GSK3923868 500 mcg | Cohort 2: GSK3923868 1000 mcg | Cohort 2: GSK3923868 3000mcg
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9
Hour (h) | 1 [1 to 2] | 1 [1 to 2] | 1 [0.8 to 1] | 1 [0.5 to 1] | 1 [0.8 to 2] | 0.75 [0.75 to 1]

21. Secondary Outcome: Part B, Cohort 3 and 4: AUC From Time Zero (Predose) to Time Tau (AUC [0-tau]) (Tau=24hours for Once a Day Dosing Regimen) of GSK3923868
Description: Blood samples were collected for measurement of plasma concentrations of GSK3923868 for PK analysis. Area under the concentration-time curve from time zero (predose) to time tau (dosing interval) was reported. Part B assessed repeat doses of study drug across two parallel cohorts (Cohorts 3 and 4).
Time Frame: Up to Day 14
Population: The analysis was performed on the PK Set that includes all randomized participants who received at least 1 dose of study intervention and had at least 1 non-missing PK assessment (NQ values were to be considered as non-missing values). Participants were analyzed according to the treatment they received. One participant was withdrawn before dosing on Day 4 and did not contribute to the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Groups:
- Cohort 3 and 4: GSK3923868 3000mcg: Healthy participants received planned repeat doses of 3000 mcg GSK3923868 daily for 14 days.
Arm/Group | Cohort 3 and 4: GSK3923868 3000mcg
Number analyzed (Participants) | 13
h*pg/mL
  Day 1 | 128045.03 (31.39)
  Day 14 (n=12): number analyzed (Participants) | 12
  Day 14 (n=12) | 144211.68 (29.45)

22. Secondary Outcome: Part B, Cohort 3 and 4: Cmax of GSK3923868
Description: Cmax was defined as the maximum concentration of drug GSK3923868 in plasma. Blood samples were collected for measurement of plasma concentrations of GSK3923868 for PK analysis. Part B assessed repeat doses of study drug across two parallel cohorts (Cohorts 3 and 4).
Time Frame: Up to Day 14
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Cohort 3 and 4: GSK3923868 3000mcg
Number analyzed (Participants) | 13
pg/mL
  Day 1 | 32342.47 (24)
  Day 14 (n=12): number analyzed (Participants) | 12
  Day 14 (n=12) | 31270.98 (26.17)

23. Secondary Outcome: Part B, Cohort 3 and 4: Tmax of GSK3923868
Description: Tmax was defined as time required to achieve Cmax for drug GSK3923868 in plasma. Blood samples were collected for measurement of plasma concentrations of GSK3923868 for PK analysis. Part B assessed repeat doses of study drug across two parallel cohorts (Cohorts 3 and 4).
Time Frame: Up to Day 14
Population: as for outcome 21
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Cohort 3 and 4: GSK3923868 3000mcg
Number analyzed (Participants) | 13
Hour (h)
  Day 1 | 0.75 [0.75 to 1]
  Day 14 (n=12): number analyzed (Participants) | 12
  Day 14 (n=12) | 1 [0.5 to 1]

24. Secondary Outcome: Part C: AUC (0-tau) (Tau=24 Hours for Once a Day Dosing Regimen) of GSK3923868
Description: Blood samples were collected for measurement of plasma concentrations of GSK3923868 for PK analysis.
Time Frame: Up to Day 7
Population: The analysis was performed on the PK Set that includes all randomized participants who received at least 1 dose of study intervention and had at least 1 non-missing PK assessment (NQ values were to be considered as non-missing values). Participants were analyzed according to the treatment they received. One participant was withdrawn before dosing on Day 7 and did not contribute to the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Groups:
- Cohort 5: GSK3923868 3000mcg: Participants with stable asthma received a planned repeat dosing of 3000 mcg GSK3923868 daily for 7 days
Arm/Group | Cohort 5: GSK3923868 3000mcg
Number analyzed (Participants) | 8
h*pg/mL
  Day 1 | 97412.11 (39.87)
  Day 7 (n=7): number analyzed (Participants) | 7
  Day 7 (n=7) | 136461.8 (24.21)

25. Secondary Outcome: Part C: Cmax of GSK3923868
Description: as for outcome 19
Time Frame: Up to Day 7
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Cohort 5: GSK3923868 3000mcg
Number analyzed (Participants) | 8
pg/mL
  Day 1 | 27799.34 (25.2)
  Day 7 (n=7): number analyzed (Participants) | 7
  Day 7 (n=7) | 35484.07 (11.97)

26. Secondary Outcome: Part C: Tmax of GSK3923868
Description: as for outcome 20
Time Frame: Up to Day 7
Population: as for outcome 24
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Cohort 5: GSK3923868 3000mcg
Number analyzed (Participants) | 8
Hour (h)
  Day 1 | 0.758 [0.5 to 1]
  Day 7 (n=7): number analyzed (Participants) | 7
  Day 7 (n=7) | 0.75 [0.75 to 1]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, SAEs and non-serious AEs were collected for Part A: Up to Day 43; for Part B: Up to Day 28 and for Part C: Up to Day 21.
Description: Safety Set comprised of all randomized participants who received at least 1 dose of study intervention.
Arm/Group | Cohort 1: Placebo | Cohort 1: GSK3923868 50 mcg | Cohort 1: GSK3923868 100 mcg | Cohort 1: GSK3923868 250mcg | Cohort 2: Placebo | Cohort 2: GSK3923868 500 mcg | Cohort 2: GSK3923868 1000 mcg | Cohort 2: GSK3923868 3000mcg | Cohort 3 and 4: Placebo | Cohort 3 and 4: GSK3923868 3000mcg | Cohort 5: Placebo | Cohort 5: GSK3923868 3000mcg
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/4 | 0/13 | 0/3 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/4 | 0/13 | 0/3 | 0/8
Other Adverse Events (participants affected / at risk) | 3/9 | 3/9 | 3/9 | 6/9 | 5/9 | 5/9 | 5/9 | 3/9 | 4/4 | 12/13 | 3/3 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Placebo (N=9) | Cohort 1: GSK3923868 50 mcg (N=9) | Cohort 1: GSK3923868 100 mcg (N=9) | Cohort 1: GSK3923868 250mcg (N=9) | Cohort 2: Placebo (N=9) | Cohort 2: GSK3923868 500 mcg (N=9) | Cohort 2: GSK3923868 1000 mcg (N=9) | Cohort 2: GSK3923868 3000mcg (N=9) | Cohort 3 and 4: Placebo (N=4) | Cohort 3 and 4: GSK3923868 3000mcg (N=13) | Cohort 5: Placebo (N=3) | Cohort 5: GSK3923868 3000mcg (N=8)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Medical device site dermatitis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase inc (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase i (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 5 (5) | 0 (0) | 7 (7)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 7 (7) | 1 (1) | 3 (3)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Product after taste (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Product taste abnormal (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT04585009/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT04585009/SAP_001.pdf